CLINICAL TRIAL: NCT02929511
Title: Influence of Reciprocating and Rotational Single-file Systems on the Postoperative Pain: A Randomized Clinical Trial.
Brief Title: Reciprocation vs Rotational Single-file Systems in Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isparta Military Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IAH-3
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2017-03

CONDITIONS: Apical Periodontitis; Assessment, Pain; Dental Pulp Necrosis
MeSH Terms: conditions — Periapical Periodontitis; Pain; Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reciproc Blue (Experimental): Endodontic treatment will be performed in teeth with necrotic pulp and periapical periodontitis. Local anaesthesia will be provided (2% Novocaine with 1:80,000 epinephrine), isolation with rubber dam and standard access cavity preparation will be done.Using 2.5 % sodium hypochlorite, canal negotiation will be done. Coronal flaring with # 2 and #3 Gates-Glidden drills will be done. The canals will be obturated with gutta-percha and epoxy resin sealer. The treatments will be carried out in single-visit. In this group, intervention will be carried out by the Reciproc motor (VDW, Germany) and Reciproc Blue single-file system (VDW, Germany). The intervention is root canal treatment with the Reciproc Blue single-file system.
  Interventions: Procedure: Reciprocating single-file system
- OneShape (Experimental): In this group, OneShape rotational single-file system (Micro Mega, France) will be used as single-file system according to the manufacturer's instruction.
  Interventions: Procedure: Rotational single-file system.
- Protaper (Active Comparator): As a control group, Protaper (Dentsply, Mailleffer, Switzerland) will be used according to the manufacturer's instruction.
  Interventions: Procedure: Active comparator Protaper multi-file system

INTERVENTIONS:
Procedure: Reciprocating single-file system — The device is moving in CW and CCW direction with different angles. It is a single-file endodontic file. The intervention is Reciproc Blue reciprocating single-file system.
  Other Names: Reciproc Blue
  Arms: Reciproc Blue
Procedure: Rotational single-file system. — The device is moving in continuous rotational. It is a single-fie endodontic file.
  Other Names: OneShape
  Arms: OneShape
Procedure: Active comparator Protaper multi-file system
  Arms: Protaper

SUMMARY:
In this study, the researchers will investigate the effect of single-file reciprocating versus single-file rotational file systems on the postoperative pain in adult patients who have necrotic pulp and apical periodontitis. The participants will be assigned by chance to separate groups that compare 2 different treatments, reciprocating single-file system (Reciproc Blue) and rotational single-file system (OneShape). As a reference, Mtwo multi-file (full-sequence) will be used.

DETAILED DESCRIPTION:
The infected root canal treatments will be performed using one-visit approach with either a reciprocating single-file system or a continuous rotational single-file system. (Reciproc Blue reciprocating single-file system vs OneShape rotational single-file system). The root canals will be completed in single-visit. The patients will record their postoperative pain during the follow-up period using a VAS scale.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have in their mandibular or maxillary molar teeth necrotic pulp and apical periodontitis.

Exclusion Criteria:

* Pregnancy, drug hypersensitivity, cardiac problems, previously performed endodontics treatment.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Pain level | 7 days.
  A VAS scale will be used for the postoperative pain level. The patients will noted their postoperative pain level according to the VAS scale during the follow-up period.

SECONDARY OUTCOMES:
Analgesic usage | 7 days.
  The patients will record the consumption of the analgesic during the 7 days of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim E YAYLALI, PhD, Principal Investigator — Devlet hastanesi
Locations (1):
- Askeri Hastane, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes